CLINICAL TRIAL: NCT07241078
Title: The Effect of WhatsApp-Based and Family-Involved Self-Management Education and Support on HbA1c, Family Support, and Self-Management in Individuals With Type 2 Diabetes
Brief Title: WhatsApp-Based and Family-Involved Diabetes Self-Management Education Study
Acronym: WAF-DSMES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Aleyna Özkan, PhD Student, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025.332.IRB2.154
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 2; Diabete Mellitus; Diabetes Education; Self-management
Keywords: diabetes; family involved; WhatsApp based; family support; HbA1c; self management; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 22 adults with type 2 diabetes and their 22 family members will receive a 12-week WhatsApp-supported, family-involved diabetes self-management education program.
  Interventions: Behavioral: WhatsApp-based Family-Involved Diabetes Self-Management Education
- Control arm (Other): 22 adults with type 2 diabetes and their 22 family members will continue standard outpatient care for 12 weeks, according to their routine clinic appointments.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: WhatsApp-based Family-Involved Diabetes Self-Management Education — Participants in the intervention group will receive a 12-week family-involved diabetes self-management education program delivered via WhatsApp. Education materials, including videos and visual guides, will be sent twice weekly (Monday and Tuesday) to both the diabetic participant and a designated family member. Participants will complete a 5-question quiz each Thursday to reinforce learning. Additionally, diabetic participants will have a weekly 10-minute phone call (Friday or Saturday) with the researcher to review progress and receive individualized feedback. Data collection will occur at baseline and at the end of the 12-week intervention using standardized forms and validated scales.
  Arms: Intervention arm
Other: Standard Care (in control arm) — Participants in the control group will continue their usual outpatient follow-up visits. This includes attending scheduled appointments with their physician and, if needed, consulting with the clinic's diabetes nurse. No additional educational intervention or structured self-management program will be provided. Data collection will occur at baseline (week 0) and at the end of week 12 using. Family members of control participants will also complete relevant forms at baseline and week 12.
  Arms: Control arm

SUMMARY:
The aim of this study is to evaluate the effects of a WhatsApp-based and family-involved self-management education program on self-management, family support, and HbA1c levels among individuals with type 2 diabetes mellitus (T2DM).

Hypotheses:

* H1: There will be a significant difference in self-management scores between the intervention group receiving the WhatsApp-based and family-involved self-management education and the control group.
* H2: There will be a significant difference in HbA1c levels between the intervention group receiving the WhatsApp-based and family-involved self-management education and the control group.
* H3: There will be a significant difference in family support scores between the intervention group receiving the WhatsApp-based and family-involved self-management education and the control group.

This randomized controlled trial will be conducted with 44 individuals diagnosed with T2DM who meet the inclusion criteria and one family member per participant (total 88 participants). Eligible patients will be randomly assigned to either the intervention or control group using a computer-generated randomization list.

Participants (people with diabetes and their family members) in the intervention group will receive a 12-week, WhatsApp-based self-management education program. Educational modules (videos, visuals, and written materials) will be shared separately with each person with diabetes and their participating family member via WhatsApp twice a week. To reinforce learning, a five-question quiz will be sent separately to both the person with diabetes and the family member every Thursday. In addition, a brief follow-up phone call (approximately 10 minutes) will be conducted once a week only with the person with diabetes to review progress and provide feedback. Data collection will occur at baseline and at the end of the 12th week.

Participants in the control group will continue their routine outpatient follow-ups for three months and complete the same measurement tools at baseline and post-intervention.

Data will be collected using the Diabetic Participant Demographic Form, Family Member Demographic Form, Diabetes Self Management Questionnaire, Hensarling's Diabetes Family Support Scale, and the Diabetes Knowledge Scale for Adults. Statistical analyses will be performed using SPSS software. Group comparisons will be analyzed with independent t-tests or Mann-Whitney U tests, and pre-post comparisons with paired t-tests or Wilcoxon tests. A significance level of p<0.05 will be used.

DETAILED DESCRIPTION:
This randomized controlled trial investigates a 12-week WhatsApp-based self-management education program for adults with type 2 diabetes mellitus (T2DM) and one designated family member per participant. The program is delivered through mobile presentations-including videos, visuals, and text-based materials-sent separately to the person with diabetes and their family member twice weekly, on Mondays and Tuesdays.

Weekly reinforcement is provided through a five-question quiz, sent individually to both participants every Thursday, and a brief (~10-minute) telephone call with the person with diabetes on Friday or Saturday, according to their preference, to review weekly progress, provide feedback, and address challenges. The intervention aims to support adherence to self-care behaviors, enhance diabetes knowledge, and strengthen family involvement.

Diabetic participants in the control group will continue their usual care, including routine physician appointments and consultations with a diabetes nurse if needed. Family members will maintain their normal daily activities without any structured intervention.

Data collection occurs at baseline and after the 12-week intervention. The study employs standardized, validated instruments including the Diabetic Participant Demographic Form, Family Member Demographic Form, Diabetes Self Management Questionnaire, Hensarling's Diabetes Family Support Scale, and the Diabetes Knowledge Scale for Adults.

Data Collection for Participants with Diabetes:

* Baseline (Week 0):

  * Diabetic Participant Demographic Form
  * Diabetes Self-Management Questionnaire
  * Hensarling's Diabetes Family Support Scale
  * Diabetes Knowledge Scale for Adults
* Post-intervention (Week 12):

  * Diabetes Self-Management Questionnaire
  * Hensarling's Diabetes Family Support Scale
  * Diabetes Knowledge Scale for Adults

Data Collection for Family Members:

* Baseline (Week 0):

  * Family Member Demographic Form
  * Diabetes Knowledge Scale for Adults
* Post-intervention (Week 12):

  * Diabetes Knowledge Scale for Adults

This study demonstrates a digitally-supported, family-involved intervention model, leveraging WhatsApp to increase accessibility, continuity, and sustainability of diabetes self-management practices. By delivering structured educational content, individualized feedback, and support from more knowledgeable family members, the program aims to enhance self-management behaviors and metabolic outcomes among adults with T2DM.

ELIGIBILITY:
Inclusion Criteria: People diagnosed with type 2 diabetes at least six months prior, receiving insulin and/or oral antidiabetic therapy, with an HbA1c value of 7% or higher, capable of communicating in Turkish, literate, and possessing the ability to use a smartphone and WhatsApp, as well as having internet access. Participants are required to agree to participate together with a family member who can provide support related to diabetes. Family members involved in the intervention are expected to be able to communicate in Turkish, literate, able to use a smartphone and WhatsApp, have internet access, and reside within reach of the participant with diabetes.

-

Exclusion Criteria: Individuals will be excluded if they have type 1 diabetes or gestational diabetes, severe cognitive impairment, advanced visual or hearing loss, any condition preventing the use of digital platforms, or communication or language barriers that would hinder participation. Family members will be excluded if they have diabetes, cognitive impairment, advanced visual or hearing loss, inability to use digital tools, or communication and language barriers.

-

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
HbA1c Level | Baseline (week 0) and 12 weeks
  HbA1c values will be obtained from participants' medical records or recent laboratory results. HbA1c reflects average blood glucose levels over the past 2-3 months. Values are reported as percentages, with higher percentages indicating poorer glycemic control.
Diabetes Self-Management | Baseline (week 0) and 12 weeks
  Measured using the Diabetes Self-Management Scale to evaluate participants' self-management behaviors. Higher scores indicate better self-management behaviors.
Family Support | Baseline (week 0) and 12 weeks
  Perceived family support in diabetes management will be assessed using Hensarling's Diabetes Family Support Scale (HDFSS). The scale includes 24 items across 4 subscales and uses a 5-point Likert response format, where higher scores indicate greater perceived family support.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Yıldız Ayvaz, Study Director — Koç University
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Results from this study will be shared with the scientific community through peer-reviewed publications.
Supporting Information: Study Protocol, CSR
Time Frame: Findings from this study are anticipated to be made available through publication within two years and will remain accessible indefinitely.
Access Criteria: Following publication, researchers working on diabetes will be able to access the study findings via the published reports.

REFERENCES:
- [Background] Walker RJ, Gebregziabher M, Martin-Harris B, Egede LE. Understanding the influence of psychological and socioeconomic factors on diabetes self-care using structured equation modeling. Patient Educ Couns. 2015 Jan;98(1):34-40. doi: 10.1016/j.pec.2014.10.002. Epub 2014 Oct 22. PMID 25455793
- [Background] Vongmany J, Luckett T, Lam L, Phillips JL. Family behaviours that have an impact on the self-management activities of adults living with Type 2 diabetes: a systematic review and meta-synthesis. Diabet Med. 2018 Feb;35(2):184-194. doi: 10.1111/dme.13547. Epub 2017 Dec 8. PMID 29150863
- [Background] Association of Diabetes Care and Education Specialists; Kolb L. An Effective Model of Diabetes Care and Education: The ADCES7 Self-Care Behaviors. Sci Diabetes Self Manag Care. 2021 Feb;47(1):30-53. doi: 10.1177/0145721720978154. PMID 34078208
- [Background] Nkhoma DE, Soko CJ, Bowrin P, Manga YB, Greenfield D, Househ M, Li Jack YC, Iqbal U. Digital interventions self-management education for type 1 and 2 diabetes: A systematic review and meta-analysis. Comput Methods Programs Biomed. 2021 Oct;210:106370. doi: 10.1016/j.cmpb.2021.106370. Epub 2021 Aug 26. PMID 34492544
- [Background] Bekele BB, Negash S, Bogale B, Tesfaye M, Getachew D, Weldekidan F, Balcha B. Effect of diabetes self-management education (DSME) on glycated hemoglobin (HbA1c) level among patients with T2DM: Systematic review and meta-analysis of randomized controlled trials. Diabetes Metab Syndr. 2021 Jan-Feb;15(1):177-185. doi: 10.1016/j.dsx.2020.12.030. Epub 2020 Dec 19. PMID 33360516
- [Background] Sacks DB, Arnold M, Bakris GL, Bruns DE, Horvath AR, Lernmark A, Metzger BE, Nathan DM, Kirkman MS. Guidelines and Recommendations for Laboratory Analysis in the Diagnosis and Management of Diabetes Mellitus. Diabetes Care. 2023 Oct 1;46(10):e151-e199. doi: 10.2337/dci23-0036. PMID 37471273